CLINICAL TRIAL: NCT00784966
Title: Pancreatic Islet Transplantation in Patients With Type 1 Diabetes Mellitus
Brief Title: Islet After Kidney Transplant for Type 1 Diabetes
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: University decision.
Sponsor: Virginia Commonwealth University (Other)
Collaborators: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VCU IRB 4196
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Islet transplantation; Type 1 Diabetes Mellitus; Kidney Transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Two weeks etanercept post islet transplant
  Interventions: Drug: etanercept
- 2 (Active Comparator): Two months etanercept treatment post islet transplant
  Interventions: Drug: etanercept

INTERVENTIONS:
Drug: etanercept — Treatment option 'A'-Two weeks treatment with etanercept. The first dose of 50mg in normal saline will be given intravenously one hour before transplant. Then 25mg will be administered subcutaneously two times a week for two weeks.
  Other Names: Enbrel
  Arms: 1
Drug: etanercept — Etanercept will be given for a total of 2 months. The first dose of 50mg in normal saline will be given intravenously one hour before transplant. Then 25mg will be administered subcutaneously two times a week for two months.
  Other Names: Enbrel
  Arms: 2

SUMMARY:
The purpose of this study is to determine if prolonged administration of the anti TNF (tumor necrosis factor)-Alpha agent etanercept is associated with enhanced graft survival in patients undergoing islet after kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes mellitus, who have a stable functioning renal transplant, are taking the appropriate maintenance immunosuppression and have no severe health problems that preclude them receiving an islet transplant will be considered for inclusion.

Exclusion Criteria:

* Have a history of or findings suggestive of unstable diabetic complications (e.g. active eye disease)
* Active infections (clinically or by laboratory testing)
* History of current malignancy or suspicion of malignancy until properly investigated and excluded
* Liver or biliary abnormalities
* Unstable cardiovascular disease
* Findings to suggest immunological sensitization or those women who have the potential to get pregnant and are not using a sufficient method of contraception

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2015-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
The functional capability of the islet allograft to normalize glucose metabolism in the absence of insulin therapy. | Outcome measures will be assessed at protocol prescribed intervals. Long term outcomes assessment will be measured at 5 years post transplant or all evidence of islet function has ceased plus six months.

SECONDARY OUTCOMES:
Reduction in insulin requirements in those patients who do not achieve insulin independence with improved metabolic control. | Outcome measures will be assessed at protocol prescribed intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian H Cotterell, M.D., Principal Investigator — Virginia Commonwealth University Health System; John N Clore, M.D., Principal Investigator — Virginia Commonwealth University Health System
Locations (1):
- Virginia Commonwealth University Health System, Richmond, Virginia, United States